CLINICAL TRIAL: NCT06117124
Title: The BoDI (Bone Density Investigation) Study: Comparing Quantitative Ultrasound and Digital X-Ray Radiogrammetry in the Investigation of Bone Density in Children with Cerebral Palsy
Brief Title: The BoDI (Bone Density Investigation) Study
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Sussex Community NHS Foundation Trust (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: 325440
Record Dates: First submitted 2023-10-24; First posted 2023-11-03 (Actual); Last update posted 2025-03-25 (Actual); Status verified 2025-03

CONDITIONS: Cerebral Palsy
MeSH Terms: conditions — Cerebral Palsy

STUDY DESIGN:
Intervention Model Description: This is a cross-sectional study whose primary objectives are to compare agreement between two bone densitometry techniques in children with cerebral Palsy, and to correlate assessments using both techniques with clinical findings.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Quantitative ultrasound (Active Comparator): Participants will undergo bone density measurement using two different modalities - quantitative ultrasound and digital x-ray radiogrammetry. Each method will be performed twice over a 12 month period, to assess changes in bone density over time.
  Interventions: Radiation: Digital X-Ray Radiogrammetry; Diagnostic Test: Quantitative Ultrasound (QUS)
- Digital x-ray radiogrammetry. (Active Comparator): Participants will undergo bone density measurement using two different modalities - quantitative ultrasound and digital x-ray radiogrammetry. Each method will be performed twice over a 12 month period, to assess changes in bone density over time.
  Interventions: Radiation: Digital X-Ray Radiogrammetry; Diagnostic Test: Quantitative Ultrasound (QUS)

INTERVENTIONS:
Radiation: Digital X-Ray Radiogrammetry — An x-ray of the left hand will be taken by a Radiographer. This will be uploaded to PACS and analysed using BoneXpert software. This calculates bone density as a 'Bone Health Index', and provides a standard deviation score for age, gender and bone age.
Diagnostic Test: Quantitative Ultrasound (QUS) — The MiniOmni Bone Densitometer will be used to measure bone density at three peripheral sites on both sides of the body (left and right): the distal radius (lower arm), mid-tibia (lower leg) and phalynx (hand). The speed of ultrasound (speed of sound) through the bone will be measured and converted to a standard deviation score.

SUMMARY:
Background:

This study involves children with cerebral palsy, a lifelong condition caused by early damage to the developing brain.

This condition is associated with impairments in mobility and motor control, eating and drinking, communication and learning, as well as other physical health difficulties. Included in these is a risk of developing osteoporosis, that is thin, weakened bones which are more prone to fracture.

Currently there is no clear guidance for how bone density should be measured or monitored in this vulnerable group of children. The recommended imaging method in children, dual energy x-ray absorptiometry (DEXA) has specific and significant limitations in children with cerebral palsy.

Aim:

This study aims to investigate two alternative methods of measuring bone density, quantitative ultrasound and digital x-ray radiogrammetry. The former uses ultrasound to measure the strength and elasticity of bone, while the latter uses hand x-rays to calculate bone density. It aims to explore the reliability, acceptability and clinical utility of both methods, as well as the correlation between the two methods. Risk factors and the clinical course of the disease will also be explored.

Method:

The study aims to recruit 70 children and young people aged 3-18 years with cerebral palsy. Participants will undergo both methods of bone density measurement twice over a 12-month period. Information on clinical risk factors and fracture rate will be taken from clinical records.

DETAILED DESCRIPTION:
Osteoporosis is a condition in which bone strength and structure is altered, so that it is more likely to break or fracture. It is a condition that has been traditionally associated with age, with women of a post-menopausal age particularly at risk. However, poor bone strength (or medically termed 'bone density') is increasingly recognised in children suffering from chronic health conditions. It is usually caused by a combination of the disease process itself, as well as the treatments and consequences of the disease.

Where childhood is usually the critical period in which bone strength is developed (and 'bone mass' accrued), these at-risk children enter adulthood with much weaker bones and at much higher ongoing risk of fracture. To minimise this risk in adulthood, the core difficulty with bone strength in childhood needs to be addressed. Of all childhood chronic health conditions, cerebral palsy is the most common condition associated with low bone density. It affects 2.7 in 1000 births and is increasing in incidence due to the increased survival of low-birth-weight infants. Low bone density is universal in children with moderate to severe Cerebral Palsy after the age of 10 years, and up to a quarter of these children will present with low-impact fractures. These are associated with pain, loss of function and quality of life, as well as significant complications, and they currently represent the most common medical problem seen in children with cerebral palsy attending residential schools.

There is currently no clear guidance for this population of at-risk children with regards to the appropriate method or timing of bone density screening. In addition, while Dual energy x-ray absorptiometry (DEXA) is currently the recommended method for measurement of bone density in children and adolescents, it has a number of limitations specifically in children with cerebral palsy. These include difficulties with accessing appropriate scanners, challenges regarding positioning and movement during scanning, and other challenges such as metallic implants from spinal and hip surgeries impacting on the ability to achieve accurate results. There is an increasing interest therefore in alternative methods of measuring bone strength in children. In 2021, a systematic review paper analysed 22 studies comparing alternative methods to DEXA in children; it concluded that quantitative ultrasound and digital x-ray radiogrammetry were both reliable methods that warrant further investigation. Of note, none of the included studies focused on children with cerebral palsy.

This study would be the first to investigate the use of these two alternative methods in children with cerebral palsy. It will address the important question of whether there is a role for these potentially more acceptable methods in screening for low bone density and predicting future fracture risk. It will also align with the research priority set by the James Lind Alliance in 2022 of managing 'distressing symptoms such as pain' in children with neurological conditions.

The aim of this study is to compare quantitative ultrasound and digital x-ray radiogrammetry as alternative and more suitable methods of bone densitometry in children with cerebral palsy.

The primary objectives of the study are:

* To compare agreement between the two densitometry techniques in children with Cerebral Palsy
* To investigate the correlation between assessments using both techniques and clinical information/ risk factors for low bone density in children with Cerebral Palsy

The secondary objectives of the study are:

* To compare bone density changes over time and identify the most appropriate timing and site of bone density screening in children with Cerebral Palsy
* To establish the risk factors associated with low bone density and pathological (low impact) fracture in this at-risk group of children
* To compare intra- and interobserver variability for both methods: that is, how consistent the results are when the investigation is performed on the same patient by the same practitioner, and on the same patient by a different practitioner.
* To compare the practicality of both methods (from the participant and practitioner viewpoint) and the cost-effectiveness of both methods
* To devise a large multi-centre trial comparing the superior of the two methods to DEXA scanning.

ELIGIBILITY:
Inclusion Criteria:

* Aged 3-18 years of age (male and female)
* Diagnosis of mild to severe cerebral palsy (Gross Motor Function Classification System Level 1 to 5)

Exclusion Criteria:

* Progressive or other neurological condition not diagnostic of Cerebral Palsy
* Previous treatment with bisphosphonates or other bone density modifying medications (aside from nutritional supplements)
* Other underlying conditions associated with low bone density e.g. malignancy or inflammatory conditions

Ages: 3 Years to 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 70 (Estimated)
Dates: Start 2025-08 (Estimated); Primary Completion 2029-01 (Estimated); Study Completion 2029-01 (Estimated)

PRIMARY OUTCOMES:
Measures taken by two densitometry techniques (quantitative ultrasound and digital x-ray radiogrammetry) | 12 months
  Level of agreement between the two techniques and correlation of both techniques with clinical findings

SECONDARY OUTCOMES:
Bone density changes over time | 12 months
  - assess bone density changes over time and identify the most appropriate timing and site of bone density screening

IPD SHARING:
Plan to Share IPD: No